CLINICAL TRIAL: NCT07086807
Title: Predictors and Impact of Total Occlusion of the Infarct-Related Coronary Artery on Short-Term Mortality in Patients With Acute Myocardial Infarction
Brief Title: Predictors and Impact of Total Occlusion of the Infarct-Related Coronary Artery on Short-Term Outcomes
Status: Completed | Type: Observational
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Nikola Kos, MD, PhD, cardiologist, University Hospital Sestre Milosrdnice
Other Study IDs: KBSestreMil
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: myocardial infarcion; infarct related artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with occluded IRA: Patients with acute occlusion (TIMI 0) of the infarct-related artery (IRA) at the time of the coronary intervention due to acute myocardial infartion
- Patients with patent IRA: Patients with acute non-occlusion (TIMI 1-3) of the infarct-related artery (IRA) at the time of the coronary intervention due to acute myocardial infartion

SUMMARY:
Aim of this study is to determine the prevalence, predictors, and impact of total occlusion of the infarct-related coronary artery (IRA) on short-term mortality.

DETAILED DESCRIPTION:
We will conduct a prospective, single-center cohort study based on a clinical registry that will include consecutive patients treated for acute myocardial infarction (AMI) with percutaneous coronary intervention (PCI) at the University Hospital Centre Sestre milosrdnice, Zagreb, Croatia, between 2011 and 2018. All patients will receive treatment in accordance with the European Society of Cardiology (ESC) guidelines current at the time. Revascularization will be performed by five experienced interventional cardiologists, each with over five years of experience and performing more than 150 PCI procedures annually. The identification of the culprit lesion will be left to the discretion of the operating physician.

Patients will be excluded if they are treated without PCI, are diagnosed with myocardial infarction with non-obstructive coronary arteries (MINOCA), or undergo surgical revascularization (coronary artery bypass grafting).

Data will be collected from the hospital electronic medical records and patient charts. Mortality data will be obtained from the Croatian National Institute of Public Health cause-of-death registry. Collected variables will include baseline demographic data, medical history, chronic pre-admission pharmacotherapy, in-hospital course, complications, and procedural characteristics. All angiograms will be re-evaluated independently by two experienced interventional cardiologists. Chronic pharmacotherapy will be considered relevant if the patient has been taking the medication for at least four weeks prior to the index event. Significant carotid artery stenosis will be defined as a luminal narrowing of more than 50%.

Patients will be divided into two groups based on the patency of the infarct-related artery (IRA): those with an occluded coronary artery (OCA group) and those with a patent coronary artery (PCA group). A patent artery will be defined as having visible antegrade flow of at least TIMI grade I distal to the culprit lesion. Occlusion will be defined as complete absence of antegrade flow beyond the site of the lesion (TIMI 0), with no visible antegrade or retrograde collateral circulation. All the patients will be pretreated with 300 mg of acetylsalicylic acid and 600 mg of clopidogrel or 180 mg of ticagrelor, depending on current guidelines.

All patients will be followed until the primary endpoint is reached or for 30 days from the index hospitalization. The primary clinical endpoint will be all-cause mortality during the follow-up period.

Statistical analysis will be performed using appropriate methods depending on data distribution. Continuous variables will be expressed as medians with interquartile ranges or as means with standard deviations, as appropriate. Normality of distribution will be assessed using the Shapiro-Wilk test. To assess statistical significance between groups, the Mann-Whitney test will be used for continuous variables, and the χ² test for discrete variables. A two-sided p-value of <0.05 will be considered statistically significant. Due to multiple comparisons, adjustment by the Benjamini-Hochberg method will be applied.

Evaluation of survival over the 30-day follow-up period will be performed using Kaplan-Meier survival curves, and the log-rank test will be used to compare survival rates between groups. Cox proportional hazards regression analysis will be used to identify independent predictors of 30-day mortality. To assess independent predictors of an occlusive type of myocardial infarction, logistic regression analysis will be employed. The statistical analysis will be performed using SPSS Version 20 (IBM SPSS Statistics, New York, USA).

ELIGIBILITY:
Inclusion Criteria:

* patients treated with PCI for AMI

Exclusion Criteria:

* treated without PCI,
* diagnosed with myocardial infarction with non-obstructive coronary arteries (MINOCA),
* underwent surgical revascularization (coronary artery bypass grafting).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with PCI for AMI at the University Hospital Centre Sestre milosrdnice, Zagreb, Croatia between 2011 and 2018.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 12 months
  Death due to all reasons in a period od 12 months after myocardial infartion

IPD SHARING:
Plan to Share IPD: No